CLINICAL TRIAL: NCT03696654
Title: Prevalence of High Blood Pressure in Paediatric Patients With Sleep Disorder Breathing. Reversibility After Treatment (The Kids TRIAL STUDY).
Brief Title: High Blood Pressure in Paediatric Patients With Sleep Disorder Breathing.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion del Hospital Nacional de Paraplejicos para la Investigacion y la Integracion (Other)
Collaborators: Hospital General Universitario de Guadalajara (Unknown); Instituto de Investigación Hospital Universitario La Paz (Other); Instituto de Investigaciones del Sueño (Unknown); Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other); Hospital General Universitario Santa Lucía (Other); Hospital Universitario Araba (Other); Hospital San Pedro de Logroño (Other)
Responsible Party: Principal Investigator, OlgaMediano, Principal Investigator, Fundacion del Hospital Nacional de Paraplejicos para la Investigacion y la Integracion
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: adm00064
Record Dates: First submitted 2018-10-03; First posted 2018-10-05 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-02

CONDITIONS: Blood Pressure; Sleep-Disordered Breathing
Keywords: high blood pressure; adenotonsillectomy; sleep-disordered breathing; sleep apnea; children; cardiovascular risk
MeSH Terms: conditions — Sleep Apnea Syndromes; Hypertension

STUDY DESIGN:
Intervention Model Description: The control system of measurements will be before and after treatment on the same group of patients (children with SDB and indication for adeno-tonsillectomy). For the analysis of the main variable (mean systolic blood pressure-BP), baseline values will be obtained through ambulatory blood pressure monitoring (ABPM) in the baseline visit. In order to evaluate the impact of treatment for SDB (adeno-tonsillar surgery) on BP, the measurement will be repeated just before the surgical intervention (ABPM) and six months after surgery (ABPM) in the same group. In this way, a control group will be available (measurements just before the surgery / control group) that will be compared with the measurements of those same patients six months after the surgery (treatment group). This measure allows having control values without preventing the treatment of any patient and without causing delays in the application of the same linked to the study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Before treatment (No Intervention)
- After treatment (Active Comparator)
  Interventions: Procedure: adenotonsillar surgery

INTERVENTIONS:
Procedure: adenotonsillar surgery — when indicated, adenotonsillar surgery for SDB treatment
  Arms: After treatment

SUMMARY:
There are data supporting a possible increase in the prevalence of High Blood Pressure (HBP) in pediatric patients with Sleep Disorder Breathing (SDB). Adeno-tonsillectomy has proven to be an effective treatment in the correction of nocturnal respiratory events in the majority of patients. Our objective is to determine the presence of HBP in pediatric patients with SDB and the impact of adenotonsillar surgery on its correction. Methodology: 286 children (4-18 years old) will be included consecutively referred for suspected SDB. Variables: a) Clinical history; b) Anthropometric variables: weight, height, body mass index, neck, hip and waist perimeter c) Chervin questionnaire d) polysomnography (PSG) for the SDB assessment and e) for the HBP evaluation, ambulatory blood pressure measurement (ABPM) will be performed during 24h. In control group (not SDB) and patients without treatment, the same tests will be repeated six months after the baseline visit. Patients with indication for medical treatment, ABPM and PSG will be performed 6 months after treatment initiation. In patients with surgery indication, ABPM will be performed just before the surgical treatment and ABPM and PSG six months after the intervention. In a subgroup of patients, it will be also assessed the presence of subclinical organic damage produced by HBP: blood markers (creatinine / glomerular filtration), urine (albuminuria / proteinuria), electrocardiogram and echocardiography (left ventricle hypertrophy).

DETAILED DESCRIPTION:
HYPOTHESIS Sleep Disorder Breathing (SDB) increase the appearance of High Blood Pressure (HBP) in pediatric patients. This HBP is reversible after treatment.

OBJECTIVES

Main goal:

1. Demonstrate how the presence of SDB is associated with an increased risk of HBP in pediatric patients. Confirm that it is reversible with the treatment.

Secondary objectives:

1. Establish the relationship between the presence of hypertension and the severity of SDB (apnea-hypopnea index-AHI, desaturation index-DI).
2. To evaluate the variability along the circadian rhythm of the HBP patterns produced in pediatric patients with SDB.
3. Establish the correlation between the diagnosis of HBP measured in the clinic and ambulatory blood pressure measurement (ABPM).
4. Assess the organic damage produced:

   1. Assess the manifestation of subclinical organic damage by means of other markers such as: blood (creatinine / glomerular filtration), urine (albuminuria / proteinuria) and echocardiography (left ventricle hypertrophy).
   2. Establish the physiopathological mechanisms involved in the HBP / SDB relationship.

Multicentre, longitudinal, prospective study with control group.

1. POPULATION TO STUDY: Children between 4 and 18 years old prospectively derived for sleep study for suspected SDB.
2. Inclusion Criteria: 1) Approval of the Ethics and Clinical Trials Committee 2) Informed consent signed by the parents and / or guardians 3) Children from 4 to 18 years old assessed consecutively due to Sleep Disorders Breathing (SDB) suspicion. Exclusion criteria: 1) Associated comorbidities: Cardiovascular (including cardiac malformation), cerebrovascular or severe unstable respiratory disease that makes it impossible to complete the studies 2) Genetic diseases 3) Children with chronic insomnia and / or depressive syndrome. 4) Children with malformation syndromes (including craniofacial malformations), Down syndrome, and neuromuscular diseases 5) previous otorhinolaryngologic surgery and / or continuous positive airway pressure (CPAP) treatment 6) Contraindication for the realization of the ABPM (arrhythmias, latex allergy or coagulation disease).
3. METHODOLOGY: All children evaluated for suspected SDB will be offered to participate in the proposed research study, once the inclusion and exclusion criteria have been reviewed. Previous informed consent of their parents, a sleep study will be carried out (complete polysomnography-PSG). The night of the sleep study will be provided to parents the Chervin questionnaire for the collection of clinical data and anthropometric measurements (weight, height; body mass index; percentiles; hip perimeter; waist circumference; neck perimeter) (V1). From the results of the sleep study four groups will be created according to the severity of the SDB measured by the apnea-hypopnea index (AHI): group I: AHI < 3 / h; Group II: AHI ≥ 3 < 5 / h; group III AHI ≥ 5 < 10 / h; Group IV: AHI ≥ 10 / h. For the study of HBP, arterial pressure will be measured in clinic and 24h ambulatory blood pressure measurement (ABPM) in a maximum time of 15 days around the completion of the sleep study (V2) (BP measures according to the regulations European 2016 collected in the study manual of procedure). All patients will be offered voluntary participation in the determination of organic subclinical damage related to HBP and pathophysiological mechanisms involved, which will include the following determinations: blood sample extraction, urine analysis, electrocardiogram and thoracic echocardiography. All organic damage tests will be carried out within a maximum period of one month around the completion of each sleep study. Once the sleep study is done, the therapeutic decision will be made in the pediatric office according to the criteria established in the regulation of sleep respiratory disorders in children SEPAR (V3) (Alonso ML et al. Arch Bronchoneumol 2011, Consensus document of the apnea-hypopnea syndrome during sleep in children). In order to evaluate the impact of treatment of SDB on HBP, measurements will be repeated after treatment (V4). In the case of patients who do not require treatment or who are referred for medical treatment tests will be repeated 6 months after the therapeutic decision making ABPM, PSG and tests of organic damage if applicable. In the case of patients referred for adenotonsillar surgery, ABPM will be repeated just before the intervention and six months after the intervention (ABPM, PSG and proof of organic damage if applicable). In this way, a control group will be available without denying treatment to any of the patients and without allowing delays in the application of the same linked with the study.

ELIGIBILITY:
Inclusion Criteria:

* Approval of the Ethics and Clinical Trials Committee
* Informed consent signed by the parents and / or guardians
* Children from 4 to 18 years old assessed consecutively due to SDB suspicion.

Exclusion Criteria:

* Associated comorbidities: Cardiovascular (including cardiac malformation), cerebrovascular or severe unstable respiratory disease that makes it impossible to complete the studies
* Genetic diseases
* Children with chronic insomnia and / or depressive syndrome
* Children with malformation syndromes (including craniofacial malformations), Down syndrome, and neuromuscular diseases
* Previous otorhinolaryngologic surgery and / or CPAP treatment
* Contraindication for the realization of the ABPM (arrhythmias, latex allergy or coagulation disease).

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 286 (Estimated)
Dates: Start 2019-02-19 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Mean systolic and diastolic blood pressure | 6 months
  Demonstrate how the presence of SDB is associated with an increased risk of HBP in pediatric patients. Confirm that it is reversible with the treatment

SECONDARY OUTCOMES:
Apnea hypopnea index | 6 months
  Establish the relationship between the presence of hypertension and the severity of SDB (apnea-hypopnea index-AHI, desaturation index-DI).
Percentage of change of mean blood pressure between day and night | 6 months
  To evaluate the variability along the circadian rhythm of the HBP patterns produced in pediatric patients with SDB
blood pressure in clinic | 6 months
  Establish the correlation between the diagnosis of HBP measured in the clinic and ambulatory blood pressure measurement (ABPM).
creatinine / glomerular filtration, albuminuria / proteinuria and left ventricle hypertrophy. | 6 months
  Assess the manifestation of subclinical organic damage by means of other markers such as: blood (creatinine / glomerular filtration), urine (albuminuria / proteinuria) and echocardiography (left ventricle hypertrophy).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario de Guadalajara, Guadalajara, Guadalajara, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Castillo-Garcia M, Solano-Perez E, Romero-Peralta S, Viejo-Ayuso ME, Silgado-Martinez L, Alvarez-Balado L, Mediano San Andres R, Resano-Barrio P, Garcia-Rio F, Cano-Pumarega I, Sanchez-de-la-Torre M, Ortigado A, Lopez-Duenas A, Fidalgo L, Rodriguez A, Mediano O, Network SS. Prevalence of High Blood Pressure in Pediatric Patients with Sleep-Disordered Breathing, Reversibility after Treatment: The KIDS TRIAL Study Protocol. Children (Basel). 2022 Nov 28;9(12):1849. doi: 10.3390/children9121849. PMID 36553294